CLINICAL TRIAL: NCT01952366
Title: Prognosis of Depression in the Elderly (PRODE)
Brief Title: Prognosis of Depression in the Elderly (PRODE). A Multicentre, Longitudinal Study of Elderly Depressed Patients.
Acronym: PRODE
Status: Completed | Type: Observational
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other); Norwegian Centre for Ageing and Health (Other); Leagacy of Josef and Haldis Andresen (Unknown); Solveig and Johan P's Foundation for Psychiatric Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: PRODE-2013
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Results first posted 2016-09-22 (Estimated); Last update posted 2023-11-27 (Actual); Status verified 2018-06

CONDITIONS: Depression; Dementia
Keywords: Aged; Depression; Cognition; Longitudinal study
MeSH Terms: conditions — Depression; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Apolipoprotein E polymorphism
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Depressed patients: Patients admitted to specialist health care service of old age psychiatry

SUMMARY:
PRODE is a Norwegian multicentre study investigating the prognosis of depression in the elderly. The study has included 169 patients who will be followed with assessments after one and three years.

The study hypothesis is that elderly patients referred to specialist health service have a poor long term prognosis.

DETAILED DESCRIPTION:
Objective: Depression in the elderly is difficult to treat and is often of chronic or recurrent nature. There is little knowledge about the course and the risk factors for recurrence of depression among elderly people in Norway. The aim of the PRODE-study is to examine the short- and long-term prognosis of elderly depressed patients who are referred for treatment in departments of old age psychiatry.

Method: PRODE is a multicentre case-control and longitudinal study of elderly (>60 years) depressed and non-depressed patients with a one and three year follow-up. Nine participating departments of old age psychiatry used the same standardized instruments to collect data of the patients on depression and other mental health issues, cognition, physical health, medications, functions in activities of daily living, quality of life and family carers' situation. The included patients and controls underwent an MRI scan of the brain according to a comprehensive protocol developed for this project. Furthermore, blood and saliva from the included patients are stored in a Biobank for analyses of pro- and anti-inflammatory cytokines and cortisol.

The study included 169 patients (December 2009-January 2013) and will include the same number of non-depressed controls.

Outcome Measures (short-term):

* Depression as measured with the Montgomery and Asberg Depression Rating Scale (MADRS), Cornell Scale for Depression in Dementia (CSDD) and Hospital Anxiety and Depression Scale (HADS), trajectories and clinical assessments.
* Function in activities of daily living

Outcome measures (long-term):

* Cognition as measured by Mini Mental State Examination (MMSE) and diagnosis of dementia.
* Depression, recurrence of depression and as measured wtih the MADRS and CSDD.
* Use of health care facilities; nursing home.
* Mortality
* Function in activities of daily living

ELIGIBILITY:
Inclusion Criteria:

* Patients with depression referred to treatment at specialist health care in Norway.
* Patients above 60 years

Exclusion Criteria:

- Demented patients with severe aphasia and patients with life threatening diseases will be excluded

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly (>60 years) depressed patients referred to treatment at specialist helth care service in Norway.
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2009-12; Primary Completion 2013-01 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geir Selbaek, MD/Ph.D, Study Director — Norwegian Centre for Ageing and Health; Tom Borza, MD/PhD cand, Principal Investigator — Innlandet Hospital Trust (Sykehuset Innlandet HF)
Locations (1):
- Innlandet Hospital Trust, Ottestad, Norway

REFERENCES:
- [Derived] Borza T, Engedal K, Bergh S, Benth JS, Selbaek G. The course of depression in late life as measured by the Montgomery and Asberg Depression Rating Scale in an observational study of hospitalized patients. BMC Psychiatry. 2015 Aug 5;15:191. doi: 10.1186/s12888-015-0577-8. PMID 26242794

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Depressed Patients
Started | 169
Completed | 138
Not Completed | 31
Not completed — Death | 22
Not completed — Withdrawal by Subject | 9

BASELINE CHARACTERISTICS:
Arm/Group | Depressed Patients
Number analyzed (Participants) | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.1 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123
  Male | 46
Region of Enrollment [Number; unit: participants]
  Norway | 169

OUTCOME MEASURES:

1. Primary Outcome: Depression
Description: Response (50% improvement on the Montgomery and Asberg Depression Rating Scale (MADRS) score) Remission (defined as score of 9 or less on the MADRS)
  The MADRS is a measurement of the severity of depression and consists of 10 items rated from 0 points (no symptoms) to 6 (severe symptoms)
Time Frame: Patients were follow during their stay in the hospital; average days of stay in hospital = 68.3 (SD=46.8)
Population: Patients with complete MADRS records
Measure: Number; unit: participants
Groups:
- Response in Depressed Patients: Number of patients admitted to specialist health care service of old age psychiatry who demonstrated a response (50% improvement of the MADRS score) during stay in the hospital.
- Remission in Depressed Patients: Number of patients admitted to specialist health care service of old age psychiatry who demonstrated a remission (MADRS score of 9 or less) by the end of their hospital stay.
Arm/Group | Response in Depressed Patients | Remission in Depressed Patients
Number analyzed (Participants) | 145 | 145
participants | 99 | 74

2. Primary Outcome: Depression
Description: Relapse/recurrence of depression
Time Frame: 1 year after inclusion to the study
Population: Inpatients
Measure: Number; unit: participants
Arm/Group | Depressed Patients
Number analyzed (Participants) | 146
participants | 48

3. Secondary Outcome: Number of Patients With a Diagnosis of Dementia
Description: One year after inclusion to the study, there will be a clinical assessment of the patient including a MMSE, if possible, and to evaluate if the patients have dementia.
Time Frame: 1 year after inclusion to the study
Measure: Count of Participants; unit: Participants
Groups:
- Patient With Dementia One Year After Inclusion to the Study: Number of patients admitted to specialist health care service of old age psychiatry who were diagnosed with dementia one year after inclusion to the study
Arm/Group | Patient With Dementia One Year After Inclusion to the Study
Number analyzed (Participants) | 146
Participants | 23

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Depressed Patients
Serious Adverse Events (participants affected / at risk) | 0/169
Other Adverse Events (participants affected / at risk) | 0/169

LIMITATIONS AND CAVEATS:
The study's recruitment is finished. Analyses are ongoing from the one-year and three-year follow-up

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No